CLINICAL TRIAL: NCT01018212
Title: Effect the Cicatrix Cream in Cutaneous Groves Treatment
Brief Title: Cicatrix Cream in Cutaneous Groves
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Fernanda Pastrana, Pediatric Hospital Juan Manuel Márquez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-0902-CU
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Cutaneous Groves
Keywords: Cutaneous Groves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Cicatrix cream
  Interventions: Other: Cicatrix cream

INTERVENTIONS:
Other: Cicatrix cream — We will be carried out the topical application of the product (Cicatrix cream) in the lesions auto administration three times a day during four months, being controlled by the specialist in months consultations.
  The dose of 0,1 ml of cream for each cm. of surface, To the patient will be explained the technique of the application.

SUMMARY:
The purpose of the study is to assess the effect of CICATRIX (Asian Gotu Kola or Pennywort) usage in the treatment of cutaneous grooves. The duration of this phase 2 clinical trial will be 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Exclusion Criteria:

* Patient that refer manifestations of high sensibility to the medication or to some of the components of the product.
* Patient that don't want to participate in the study.
* Patient not very cooperative.
* Responsible family not very cooperative.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
They are the cutaneous grooves, being Observed the reduction of the number of the lesions monthly. | 4 month

SECONDARY OUTCOMES:
Extension of the groves and the reduction of these expressed in centimetres | 4 months
Adverse effects | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Pastrana, MD, Principal Investigator — Pediatric Hospital Juan Manuel Marquez
Locations (1):
- Pediatric Hospital Juan Manuel Marquez, Havana, La Habana, Cuba